CLINICAL TRIAL: NCT00106847
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Infliximab Induction Therapy Followed by Multiple Regimens of Maintenance InfliximabTherapy in Patients With Plaque-Type Psoriasis
Brief Title: A Study of the Safety and Effectiveness of Infliximab in Patients With Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005290
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Psoriasis; Parapsoriasis
Keywords: plaque-type psoriasis; psoriasis; drug safety; drug efficacy; maintenance therapy; induction therapy; remicade
MeSH Terms: conditions — Psoriasis; Parapsoriasis | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of scheduled and as needed treatment of psoriasis with infliximab. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
This is a phase III, multicenter, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled trial evaluating the effectiveness and safety of scheduled and as needed treatment with infliximab in patients with plaque-type psoriasis. This study will also help determine the way to use infliximab in treating patients with psoriasis.

Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures.

Patients will receive infusions of either placebo, 3mg/kg or 5 mg/kg infliximab (Remicade) at weeks 0, 2, 6 14, 18, 22, 26, 30, 34, 38, 42 and 46. Patients receive either 3mg/kg, 5 mg/kg or placebo infusions at week 0, 2, and 6. The 3mg/kg and 5 mg/kg infliximab groups then receive either every 8 week infusions or infusions as needed when their psoriasis is less than 75% improved from baseline. The placebo patients begin infliximab at week 16, 18 and 22 followed by every 8 week infusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of plaque-type psoriasis for at least 6 months
* Patients with plaque-type psoriasis covering at least 10% of the body

Exclusion Criteria:

* Patients with nonplaque forms of psoriasis
* Patients who have current drug-induced psoriasis
* Patients who are pregnant, nursing, or planning pregnancy (both men and women) within 18 months of enrollment
* Patients who had any previous treatment with infliximab or any therapeutic agent targeted at reducing tumor necrosis factor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2003-01; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve greater or equal to 75% improvement in Psoriasis Area and Severity Index (PASI) from baseline at week 10.

SECONDARY OUTCOMES:
Improvement from baseline in Psoriasis Area and Severity Index response between weeks 16 and 30. Change in Dermatology Life Quality Index from baseline at week 10. Patients with a Physician's Global Assessment score of clear or excellent at week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Menter A, Feldman SR, Weinstein GD, Papp K, Evans R, Guzzo C, Li S, Dooley LT, Arnold C, Gottlieb AB. A randomized comparison of continuous vs. intermittent infliximab maintenance regimens over 1 year in the treatment of moderate-to-severe plaque psoriasis. J Am Acad Dermatol. 2007 Jan;56(1):31.e1-15. doi: 10.1016/j.jaad.2006.07.017. Epub 2006 Sep 6. PMID 17097378
- See also: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of Infliximab Induction Therapy Followed by Multiple Regimens of Maintenance Infliximab Therapy in Subjects with Plaque-type Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=160&filename=CR005290_CSR.pdf